CLINICAL TRIAL: NCT02889419
Title: Benefits Evaluation of Selfia® Adapted Underwear for Multiple Sclerosis Patients With Severe to Moderate Handicap Performing Self-catheterization : a Multicenter, Prospective, Uncontrolled and Before/After Study.
Brief Title: Benefits Evaluation of Selfia® Adapted Underwear for MS Patients Performing Self-catheterization
Acronym: KML
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC-P0045
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Disability; Underwear; Urinary catheter; Self-catheterisation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation of underwear Selfia® (Experimental): Every patient is his own control.
  Interventions: Device: Evaluation of underwear Selfia®

INTERVENTIONS:
Device: Evaluation of underwear Selfia® — Patients are evaluated for a week using their usual underwear for the realization of SC. At the end of the week, they receive Selfia ® adaptated underwear and they use it for one week for a new evaluation. Finally, underwear will be given to patients and during follow-up consultations in routine at 6 months and 1 year, he will be asked if they reused or bought underwear.

SUMMARY:
KML is a multicenter, prospective, uncontrolled and before/after study. The study aims to estimate if the use of Selfia ® adapted underwear reduces the necessary duration for the realization of self-catheterisation (SC) for patients affected by multiple sclerosis with severe to moderate disability.

Secondly, the study aims to :

* Estimate the effect of underwear on quality of life, tiredness linked to the act, comfort in the realization of SC, complications with SC, third party intervention ;
* Collect patients' opinion on the use of the underwear SELFIA ® at the end of the 2nd week of evaluation ;
* Measure if the patient reused underwear and if he bought it at 6 months and at 1 year

DETAILED DESCRIPTION:
Bladder-sphincter disorders affect 80 % of the patients suffering from multiple sclerosis (MS) after 10 years of evolution and urinary self-catheterization (SC) are part of the therapeutic arsenal.

SC involves different steps: the preparation of the material, the undressing, the transfer on toilets, the technical gesture and the dressing. Recommendations of good practice of SC of the French Society of Physical Medicine and Rehabilitation evoke the necessity to adapt the wardrobe but without precision on the definition of this adaptation.

Adapted underwear exists for patients with a disability and is accessible for the general public. However, no clinical trial has ever evaluated their real practical interest for disabled patients realizing SC.

These undergarments, according to our experience, are very ingenious and would bring a real comfort in everyday life from patients with a disability.

In case of SC, this underwear would facilitate and shorten the time dedicated to this technique, especially as SC are realized on average 6 times a day for patients already affected in their movements because of their initial handicap.

The adapted underwear could bring an ease and a speed of dressing / undressing, allow an easier and faster access to the urinary meatus and a limitation of manipulations and mobilizations of the patient allowing an energy saving.

Moreover, disabled patients request concrete advice from health professionals on everyday life problems such as dressing / undressing. Therefore it seemed interesting to estimate the benefits of using adapted underwear for the realization of SC for patients affected by MS with severe to moderate disability (EDSS 6 - 7.5) affecting everyday life activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple sclerosis (MS) according to McDonald criteria
* At least 18 years old
* Self-catheterization for at least 3 months
* Expended Disability Status Scale (EDSS) between 6.0 and 7.5
* Informed consent
* Coverage of the social insurance

Exclusion Criteria:

* MS relapse in the previous month
* Patient hospitalized in short stay or aftercare departments, no matter the reason
* Morbid obesity (BMI superior to 35)
* Understanding disorders preventing an informed consent
* EDSS inferior to 6.0 or superior to 7.5
* Patient with home bladder catheter
* No capacity to provide a self-catheterisation
* Age under 18 years
* Pregnant or breast-feeding woman
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Average time spend for the realization of a self-catheterisation, from undressing to dressing, measured by a chronometer provided to the patient | 17 days

SECONDARY OUTCOMES:
Measure of the quality of life | 17 days
  Specific scale adapted for the studied population: Qualiveen (self-questionnaire for MS patients with urinary disorders)
Measure of fatigue for every SC | 17 days
  EVA scale
Comfort linked to SC | 17 days
  EVA scale for pain linked to undressing / dressing
Consequences from SC complications | 17 days
  Number of bleeding, EVA scale for the pain linked to the introduction / withdraw of the urinary catheter,
Number of documented urinary infections | 17 days
Number of self-catheterisation or hetero-catheterisation per day | 17 days
Opinion of the patient (favorable/non favorable) on the use of underwear Selfia ® | at 6 months and at 1 year
Re-use (yes/no) of underwear with or without purchase (yes/no) | at 6 months and at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Cattoir-Vue, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (6):
- France (6):
  - Groupement des Hôpitaux de l'Institut Catholique de Lille, Lomme, Hauts-de-France
  - Clinique Saint-Augustin, Bordeaux
  - Hôpital Swynghedauw - CHRU de Lille, Lille
  - Cabinet médical de Neurologie, Lyon
  - Hôpital Saint-Jacques - CHU Nantes, Nantes
  - Pôle MPR Saint Hélier, Rennes

IPD SHARING:
Plan to Share IPD: No